CLINICAL TRIAL: NCT03665129
Title: A Phase I Study of the Anti-C5aR, IPH5401, in Combination With the Anti-PD-L1, Durvalumab, in Patients With Selected Advanced Solid Tumors
Brief Title: IPH5401 (Anti-C5aR) in Combination With Durvalumab in Patients With Advanced Solid Tumors
Acronym: STELLAR-001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: early termination
Sponsor: Innate Pharma (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IPH5401-101
Record Dates: First submitted 2018-09-01; First posted 2018-09-11 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — avdoralimab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose escalation (Experimental): IPH5401 at different doses and schedule + Durvalumab
  Interventions: Biological: IPH5401 and Durvalumab
- Cohort expansion NSCLC anti-PD-(L)1 pretreated (Experimental): IPH5401 at recommended dose and schedule + Durvalumab in NSCLC anti-PD-(L)1 pretreated patients
  Interventions: Biological: IPH5401 and Durvalumab
- Cohort expansion HCC anti-PD-(L)1 naive (Experimental): IPH5401 at recommended dose and schedule + Durvalumab in HCC anti-PD-(L)1 naive patients
  Interventions: Biological: IPH5401 and Durvalumab
- Cohort expansion HCC anti-PD-(L)1 pretreated (Experimental): IPH5401 at recommended dose and schedule + Durvalumab in HCC anti-PD-(L)1 pretreated patients
  Interventions: Biological: IPH5401 and Durvalumab

INTERVENTIONS:
Biological: IPH5401 and Durvalumab — IPH5401 and durvalumab

SUMMARY:
This is a multicenter, open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability, antitumor activity of IPH5401 (anti C5aR) in combination with Durvalumab (MEDI4736) in Adult Subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced and/or metastatic histologically solid tumors with evidence of active disease, who have been treated with a minimum of one line of systemic therapy in the metastatic setting, and in expansion part, no more than two prior systemic therapies.
2. At least 18 years of age.
3. ECOG performance status of ≤1.
4. Adequate organ function

Exclusion Criteria:

1. For patients with Non Small Cell Lung Cancer (NSCLC):

   a. Known actionable mutation or rearrangement (including but not limited to the epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) gene rearrangements, ROS-1 alterations or BRAF mutations)
2. For patient with Hepatocellular carcinoma (HCC):

   1. Hepatic encephalopathy in the past 12 months.
   2. Ascites that requires repeated paracentesis in the past 2 months.
   3. Main portal vein thrombosis.
   4. Active or prior history of gastrointestinal bleeding in the past 12 months.
   5. Prior hepatic transplantation.
3. Patients with known spinal cord compression.
4. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of Drug Limited Toxicities (DLTs) | From Time of First dose assessed up to 6 weeks
  To assess the occurrence of Drug Limited Toxicities (DLTs)
Adverse events (AEs) | From screening visit up to 30 days after the last dose of study medication
  To evaluate the safety profile

SECONDARY OUTCOMES:
Objective Response Rate | up to 12 months
  Rate of patients in complete or partial response according to RECIST 1.1
Duration of Response | 2 years and 9 months
  duration between the complete or partial response and the first documented progression
Progression Free Survival | 2 years and 9 months
  time between the start of treatment and the first documented progression or death

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
- France (7):
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Hôpital de la Timone- AP-HM, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Centre Hospitalier Universitaire- Hôpital Nord Laennec, Nantes
  - Centre Eugène Marquis, Rennes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No